CLINICAL TRIAL: NCT00047567
Title: Open-label Adjunctive Zonisamide for Bipolar Disorder
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Elan Pharmaceuticals (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ELN-345-509
Record Dates: First submitted 2002-10-08; First posted 2002-10-10 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Bipolar Disorders
Keywords: ZONISAMIDE; BIPOLAR
MeSH Terms: conditions — Bipolar Disorder | interventions — Zonisamide

INTERVENTIONS:
Drug: zonisamide

SUMMARY:
To study the safety and efficacy of zonisamide as adjunctive therapy for children and adolescents with bipolar I or II disorder.

ELIGIBILITY:
* Bipolar I/II
* Average intelligence
* Taking at least one, but no more than two mood stabilizers

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20
Dates: Start 2002-07; Study Completion 2002-07